CLINICAL TRIAL: NCT05114811
Title: Effects of Perineal Massage During Pregnancy on Women's Health
Brief Title: Effects of Perineal Massage (PERMAS)
Acronym: PERMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Raquel Leirós-Rodríguez, Ph.D. Assistant Professor, Universidad de León
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OBST2021001
Record Dates: First submitted 2021-10-26; First posted 2021-11-10 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Musculoskeletal Manipulations; Primary Prevention; Obstetric Labor Complications; Physical Therapy Modalities
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis was carried out by an investigator blinded to experimental groups (unaware of the meaning of codification of the database of the three sample subgroups).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapist massage (Experimental): Perineal massage was applied by a physiotherapist expert in urogynecology and obstetrics during a total of 6 to 10 sessions (from 34th gestation week until delivery) of 30 minutes each on a weekly basis.
  Interventions: Procedure: Physiotherapist perineal massage: manual and instrumental (with EPI-NO)
- Self-massage intervention (Experimental): Self-massage group received permanent instructions on perineal massage during pregnancy: it should be applied at least twice a week (on alternate days) during 10 minutes using a water-based lubricant from the 34th gestation week until delivery.
  Interventions: Procedure: Self-provided perineal massage
- Control (No Intervention): Group receiving standard obstetric care (consultation and check-ups with the gynaecologist and midwife). No contact with the research physiotherapists.

INTERVENTIONS:
Procedure: Self-provided perineal massage — External massage should be applied with pump of the perineum central core. Internal massage should be applied intracavitary with longitudinal glides, myofascial trigger points of pelvic diaphragm and streching.
  Arms: Self-massage intervention
Procedure: Physiotherapist perineal massage: manual and instrumental (with EPI-NO) — The treatment sequence included external massage with two manouvres: vulvar drainage and pump of the perineum central core. Intracavitary techniques were then applied through three maneuvers: massage with longitudinal glides, myofascial trigger points of pelvic diaphragm and streching.
  After this, instrumental massage was applied with the EPI-NO® device.
  Arms: Physiotherapist massage

SUMMARY:
Perineal massage increases elasticity of myofascial perineal tissue and decreases the burning and perineal pain during labour, thus optimizing child birth, although an application protocol has not been standardized yet. The objective of this non-randomized controlled trial is to determine the efficiency of massage in perineal tear and urinary incontinence prevention and identification of possible differences in massage application. The sample target is to exceed 75 women analysed between January and May 2020. The interventions include: (a) perineal massage and EPI-NO® device group, applied by an expert physiotherapist; (b) self-massage group, where women were instructed to apply perineal massage in domestic household; and (c) a control group, which received ordinary obstetric attention.

Approval for the study was obtained through the Ethics Committee of the University of Leon (code: ETICA-ULE-021-2018). All participants signed an informed consent form, in accordance with the Declaration of Helsinki (rev. 2013), and had the option to revoke their participation in the study at any time. Ethical regulations were respected as well as the Spanish Law for Protection Data Organic Law and for Biomedical Research in Human Participants.

Data collection took place during an evaluation session on the fifth- or sixth- postpartum week through a self-reported form where participants registered the characteristics of delivery (gestation week, baby's weight, duration and posture of delivery, tear, episiotomy, use of equipment and/or analgesia). The form also included a question on intensity of perineal pain at the time of evaluation (quantified by visual analogue scale) and and urinary incontinence incidence through ICIQ-SF (punctuation higher than 0) and description (quantity of loss of urine and how this affects to their daily life), identified on the items included on the questionnaire.

DETAILED DESCRIPTION:
This non-randomized controlled trial has the sample target of 75 women analysed, at least, between January and May 2020.

The following inclusion criteria were defined to participate in the study: (a) women between 18 and 40 years of age; (b) full term delivery (37th week or more); (c) single gestation and with cephalic presentation; (d) pregnancy with no complications, nor added risks during gestation; (e) no participation in any other psychoprophylaxis intervention; (f) deliver at the Hospital Nuestra Señora de Sonsoles (Spain). The following exclusion criteria were simultaneously defined: (a) any contraindication for perineal massage and/or vaginal delivery; (b) medical diagnosis of any urogynecologi-cal pathology previous to gestation process; (c) any records of cesarean delivery and/or history of perineal injury and/or urinary incontinence; (d) not giving informed consent of participation in the study or lack of attendance to every programmed intervention and/or evaluation session.

Approval for the study was obtained through the Ethics Committee of the University of Leon, Spain (code: ETICA-ULE-021-2018). All participants signed an informed consent form, in accordance with the Declaration of Helsinki (rev. 2013), and had the option to revoke their participation in the study at any time. Ethical regulations were respected as well as the Spanish Law for Protection Data Organic Law and for Biomedical Research in Human Participants.

Methodology The interventions include: (a) perineal massage and EPI-NO® device group, applied by an expert physiotherapist; (b) self-massage group, where women were instructed to apply perineal massage in domestic household; and (c) a control group, which received ordinary obstetric attention. Groups were not randomized since the priority was the wellbeing of the pregnant par-ticipant and were assigned according to the participant's preferences (attendance at the medical centre for physiotherapy treatment, self-massage at home or attendance at childbirth preparation sessions only).

Data collection took place during an evaluation session on the fifth- or sixth- postpartum week through a self-reported form where participants registered the characteristics of delivery (gestation week, baby's weight, duration and posture of de-livery, tear, episiotomy, use of equipment and/or analgesia). The form also included a question on intensity of perineal pain at the time of evaluation (quantified by visual analogue scale).

Perineal self-massage intervention Self-massage group received permanent instructions on perineal massage during pregnancy: it should be applied at least twice a week (on alternate days) during 10 minutes using a water-based lubricant from the 34th gestation week until delivery. The position during self-massage should be comfortable and relaxed (recommended: lying face up or semi-seated position). External massage should be applied in semicircles (towards the medial) on both sides of the vaginal vestibule and by 'pumping' (rhyth-mically pressing and releasing) on the central core of the perineum. Internal massage should be applied intracavitary with the thumb by dorso-central glides on both vaginal lateral walls (gliding on the introitus vaginae from 8 to 11 and from 4 to 1 clockwise until tissue relaxation). Then, with the help of the index finger, identify tenser areas on the vaginal walls (such as thin strings) that could be gently pressed or rubbed and then wait for relaxation. Finally, apply tissue stretching technique by clamp traction with one intracavitary finger and other external finger until tension or discomfort, hold the position until relief and then without releasing, apply traction again. This latter tech-nique should be repeated three times on both sides (gliding on the introitus vaginae from 11 to 1 clockwise). Participants in the self-massage group received exhaustive in-formation on massage application and filled in a daily register to check on their ad-herence to guidelines given and were also checked weekly (at consultation in person or by phone).

Perineal massage intervention Perineal massage was applied by a physiotherapist expert in urogynecology and obstetrics during a total of 6 to 10 sessions (from 34th gestation week until delivery) of 30 minutes each on a weekly basis. The position of the pregnant participant is semi-seated, with her back against the stretcher and the legs on the stretchers' legs. A water-based lubricant was used for massage.

The treatment sequence included external massage with two manouvres: vulvar drainage and pump of the perineum central core. Drainage is a semicircular applica-tion with two or three fingers towards the medial on both sides of the vaginal vesti-bule, 15 semicircles on each side, in 3 series of 5 repetitions and moving forward in an-teroposterior direction. In case of identification of vulvar edema, there should be as many applications as needed. Pumps is a series of rhythmical pressures with one or two fingers (3 series of 5 repetitions, that is, 15 pumps in total). In case of muscular edema or hypertone, as many pumps as needed should be applied until normalization of tissue.

Intracavitary techniques were then applied through three maneuvers. First, mas-sage with longitudinal glides on the ani levator muscles, on both lateral walls of the vagina in anteroposterior direction (following the track of the ischiopubian branches) with the second and third fingers. There were 3 series of 5 glides on both sides, in-creasing its number until normalization of tissue. Second, application of treatment of myofascial trigger points of pelvic diaphragm identified by tense bands or active points that provoked referred pain recognizable to the patient and/or response to local spasm. In such cases, manual technique involves inhibition by pressure and/or friction until normalization of tissue and disappearance of associated symptomatology. Finally, application of manual stretches on both sides of the vagina (on the area coinciding with a future possibility of lateromedial episiotomy). The stretching was applied in three stages, moving progressively, according to the sensations of the pregnant partic-ipant and the elasticity of the perineal muscles.

After application of manual techniques, instrumental massage was applied with the EPI-NO® device. First, the device should be introduced deflated and once placed in the vagina, slowly inflated until finding the first barrier, where the pregnant partici-pant manifests sensation of stretching (never discomforting nor painful). Inflation volume was held until the pregnant participant noted her sensation of stretching di-minished, then the ball was slowly inflated again until meeting another stretching bar-rier. Three barriers should be met, and the device should be moved gently in the search for stretching barriers and local massage.

Finally, an external manual technique was applied to relax the perineal area through perineal global pumping by contacting with the first phalanx of the four last fingers of the hand (with fist closed) on the vulvar area. 3 series of 5 pumps were ap-plied.

Safety considerations None of the interventions and assessment tools used (applied as described and as recommended in the available literature) have shown adverse effects after application.

Follow-up The research protocol does not include follow-up for data collection. However, the women participants will be able to go to the physiotherapist who recruited the participants, who applied the different interventions and who collected the information analysed through direct consultation in the public health centre where it is expected that she will continue to work.

ELIGIBILITY:
Inclusion Criteria:

* Full term delivery (37th week or more).
* Single gestation and with cephalic presentation.
* Pregnancy with no complications, nor added risks during gestation.
* No participation in any other psychoprophylaxis intervention.
* Deliver at the Hospital Nuestra Señora de Sonsoles (Spain).

Exclusion Criteria:

* Any contraindication for perineal massage and/or vaginal delivery.
* Medical diagnosis of any urogynecologi-cal pathology previous to gestation process.
* Any records of cesarean delivery and/or history of perineal injury and/or urinary incontinence.
* Not giving informed consent of participation in the study or lack of attendance to every programmed intervention and/or evaluation session.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Gestation week | Post-test: fifth- or sixth- postpartum week
  Number of the gestational week in which the birth took place.
Urinary incontinence incidence | Post-test: fifth- or sixth- postpartum week
  International Consultation on Incontinence Questionnaire-Short Form
Baby's weight | Post-test: fifth- or sixth- postpartum week
  Baby's weight in kilograms at birth
Duration of delivery | Post-test: fifth- or sixth- postpartum week
  Duration of labour (in hours) from the onset of contractions to the delivery of the placenta
Posture of delivery | Post-test: fifth- or sixth- postpartum week
  Recording the mother's posture during the second stage of labour: lithotomy, lying on the side, sitting, squatting or on all fours.
Perineal tear | Post-test: fifth- or sixth- postpartum week
  Record of whether perineal tearing occurred during delivery and, if so, its severity (types: I, IIa, IIb or III).
Episiotomy | Post-test: fifth- or sixth- postpartum week
  Record of whether episiotomy was performed (or not) during delivery.
Use of equipment | Post-test: fifth- or sixth- postpartum week
  Record whether delivery instruments were used during delivery: no instruments, vacuum extraction or forceps.
Analgesia | Post-test: fifth- or sixth- postpartum week
  Record whether pharmacological analgesia was used during labour: no analgesia, epidural analgesia, spinal analgesia or local perineal analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias de la Salud, Ponferrada, León, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication of two scientific articles describing the procedure and publicly disclosing the results obtained. No individual data of any of the patients or images related to them will be disclosed.
Supporting Information: Study Protocol, ICF
Time Frame: Between 2021 and 2022.
Access Criteria: The data presented in this study are available on request from the corresponding author of the articles published.

REFERENCES:
- [Background] Ochandorena-Acha M, Noell-Boix R, Yildirim M, Cazorla-Sanchez M, Iriondo-Sanz M, Troyano-Martos MJ, Casas-Baroy JC. Experiences and coping strategies of preterm infants' parents and parental competences after early physiotherapy intervention: qualitative study. Physiother Theory Pract. 2022 Sep;38(9):1174-1187. doi: 10.1080/09593985.2020.1818339. Epub 2020 Sep 7. PMID 32892686
- [Background] Van Kampen M, Devoogdt N, De Groef A, Gielen A, Geraerts I. The efficacy of physiotherapy for the prevention and treatment of prenatal symptoms: a systematic review. Int Urogynecol J. 2015 Nov;26(11):1575-86. doi: 10.1007/s00192-015-2684-y. Epub 2015 Mar 31. PMID 25822028
- [Background] Ray-Griffith SL, Wendel MP, Stowe ZN, Magann EF. Chronic pain during pregnancy: a review of the literature. Int J Womens Health. 2018 Apr 9;10:153-164. doi: 10.2147/IJWH.S151845. eCollection 2018. PMID 29692634
- [Background] Gallo RBS, Santana LS, Marcolin AC, Duarte G, Quintana SM. Sequential application of non-pharmacological interventions reduces the severity of labour pain, delays use of pharmacological analgesia, and improves some obstetric outcomes: a randomised trial. J Physiother. 2018 Jan;64(1):33-40. doi: 10.1016/j.jphys.2017.11.014. Epub 2017 Dec 27. PMID 29289579
- [Background] Taavoni S, Abdolahian S, Haghani H, Neysani L. Effect of birth ball usage on pain in the active phase of labor: a randomized controlled trial. J Midwifery Womens Health. 2011 Mar-Apr;56(2):137-40. doi: 10.1111/j.1542-2011.2010.00013.x. Epub 2011 Feb 28. PMID 21429078
- [Background] Badaoui A, Kassm SA, Naja W. Fear and Anxiety Disorders Related to Childbirth: Epidemiological and Therapeutic Issues. Curr Psychiatry Rep. 2019 Mar 12;21(4):27. doi: 10.1007/s11920-019-1010-7. PMID 30868272
- [Background] Airo Toivanen R, Korja R, Saisto T, Rouhe H, Muotka J, Salmela-Aro K. Changes in emotions and personal goals in primiparous pregnant women during group intervention for fear of childbirth. J Reprod Infant Psychol. 2018 Sep;36(4):363-380. doi: 10.1080/02646838.2018.1462477. Epub 2018 May 7. PMID 29733686
- [Background] Dieb AS, Shoab AY, Nabil H, Gabr A, Abdallah AA, Shaban MM, Attia AH. Perineal massage and training reduce perineal trauma in pregnant women older than 35 years: a randomized controlled trial. Int Urogynecol J. 2020 Mar;31(3):613-619. doi: 10.1007/s00192-019-03937-6. Epub 2019 Apr 2. PMID 30941442
- [Background] Shahoei R, Zaheri F, Nasab LH, Ranaei F. The effect of perineal massage during the second stage of birth on nulliparous women perineal: A randomization clinical trial. Electron Physician. 2017 Oct 25;9(10):5588-5595. doi: 10.19082/5588. eCollection 2017 Oct. PMID 29238501
- [Background] Schreiner L, Crivelatti I, de Oliveira JM, Nygaard CC, Dos Santos TG. Systematic review of pelvic floor interventions during pregnancy. Int J Gynaecol Obstet. 2018 Oct;143(1):10-18. doi: 10.1002/ijgo.12513. Epub 2018 May 18. PMID 29705985
- [Background] Beckmann MM, Stock OM. Antenatal perineal massage for reducing perineal trauma. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD005123. doi: 10.1002/14651858.CD005123.pub3. PMID 23633325
- [Background] Romina S, Ramezani F, Falah N, Mafi M, Ranjkesh F. Effect of Perineal Massage with Ostrich Oil on the Episiotomy and Lacerations in Nulliparous Women: A Randomized Controlled Clinical Trial. Iran J Nurs Midwifery Res. 2020 Feb 24;25(2):134-138. doi: 10.4103/ijnmr.IJNMR_76_19. eCollection 2020 Mar-Apr. PMID 32195159